CLINICAL TRIAL: NCT02972307
Title: The Extent to Which Caregivers Enhance the Wheelchair Skills of Powered Wheelchair Users: a Descriptive Cross-sectional Study
Brief Title: Caregiver-aided Powered Wheelchair Skills
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lee Kirby, Physician, Nova Scotia Health Authority
Other Study IDs: 1020645
Record Dates: First submitted 2016-11-18; First posted 2016-11-23 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Caregivers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- caregiver: dyad of caregiver and the wheelchair user to whom they provide care
  Interventions: Other: wheelchair skills

INTERVENTIONS:
Other: wheelchair skills — the extent to which caregivers enhance the wheelchair skills of powered wheelchair users

SUMMARY:
There has been only minimal research on wheelchair skills by the caregivers of manual or powered wheelchair. There are no published data on the extent to which caregivers can enhance the mobility of powered wheelchair users. The primary objective of this study is to test the hypothesis that caregivers enhance the wheelchair skills capacity, confidence and performance of the powered wheelchair users to whom they provide assistance. Our secondary objective is to add to the literature on the measurement properties of the wheelchair skills test (questionnaire and capability version) for powered wheelchair users and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* able to communicate in English and/or French (depending upon the site)
* live within 50 km of the research centre
* be willing to participate (as evidenced by completion of the assessment)
* be able to set a scheduled time for the study visit when both the caregiver and wheelchair user will be present and provide informed consent

Caregivers:

* must be an unpaid caregiver (e.g. a family member or friend)
* spend an average total of at least 2 hours per week with the powered wheelchair user that includes powered wheelchair mobility.

Wheelchair user:

* must have his/her own powered wheelchair
* use the powered wheelchair for at least 6 hours per week
* have a caregiver who spends an average total of at least 2 hours per week with the powered wheelchair user that includes powered wheelchair mobility.

Exclusion Criteria:

* have unstable medical conditions (e.g. angina, seizures) that might make the use of a powered wheelchair dangerous
* emotional problems (e.g. severe anxiety, depression) that might make participation unsafe or unpleasant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: dyads of caregivers and the wheelchair users to whom they provide care
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Wheelchair Skills Test (WST) | one day
  Objective (WST) and Questionnaire (WST-Q) versions

SECONDARY OUTCOMES:
Questionnaire | one day
  Qualitative open ended questions on wheelchair skills

CONTACTS AND LOCATIONS:
Overall Officials: Lee Kirby, MD, FRCPC, Principal Investigator — Dalhousie University, Nova Scotia Health Authority
Locations (1):
- Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kirby RL, Rushton PW, Routhier F, Demers L, Titus L, Miller-Polgar J, Smith C, McAllister M, Theriault C, Matheson K, Parker K, Sawatzky B, Labbe D, Miller WC. Extent to Which Caregivers Enhance the Wheelchair Skills Capacity and Confidence of Power Wheelchair Users: A Cross-Sectional Study. Arch Phys Med Rehabil. 2018 Jul;99(7):1295-1302.e9. doi: 10.1016/j.apmr.2017.11.014. Epub 2018 Jan 3. PMID 29305847